CLINICAL TRIAL: NCT00979680
Title: Phase II Trial Comparing Two Neoadjuvant Treatments in Patients With Ultra-low Rectal Cancer: High-dose Radiotherapy Versus Radio-chemotherapy
Brief Title: Sphincter-preserving Surgery After Preoperative Treatment of Ultra-low Rectal Carcinoma
Acronym: GRECCAR1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Pr Philippe Rouanet, CRLC Val d'Aurelle
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBR-2001
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Rectal Cancer
Keywords: sphincter preservation; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-dose Radiotherapy (Active Comparator)
  Interventions: Radiation: High-Dose radiotherapy
- Chemo-radiotherapy (Active Comparator)
  Interventions: Radiation: Chemo-radiotherapy

INTERVENTIONS:
Radiation: High-Dose radiotherapy — Preoperative radiotherapy of 45 Gy/25 fractions of 1.8 Gy through three fields was delivered to the pelvis over 5 weeks, followed by a 18 Gy/10 fraction boost to the primary tumor over 2 weeks.
  Other Names: HDRT
  Arms: High-dose Radiotherapy
Radiation: Chemo-radiotherapy — Chemotherapy (5-fluorouracil, 200 mg per square meter of body-surface area per day) was delivered over 5 weeks concurrently with the pelvic radiotherapy.
  Other Names: CTRT
  Arms: Chemo-radiotherapy

SUMMARY:
This phase III trial included patients with low rectal adenocarcinoma which initially required APR, with a mean clinical distance between the tumor inferior pole and the levator ani of 0.5 cm. Patients were randomly assigned to receive high-dose radiation (45 + 18 Gy) or radiochemotherapy (45 Gy + 5FU continuous infusion). The surgical decision was based on the tumor status at surgery. All surgeons used a homogenous SSR technique such as intersphincteric resection. The primary endpoint was the SSR rate.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of ultra-low rectum at high risk of abdomino-périneal amputation
* Tumor classified as EER UT2-UT3, whatever the nodal status
* pathological confirmation of rectal adenocarcinoma without evidence of distant metastasis (M0), T2 or T3 resectable tumors without striated sphincter involvement and with the inferior margin of the tumor located less than 2 cm from the upper part of the levator ani.
* Age 18 years or older
* Informed and written consent

Exclusion Criteria:

* T1
* T4 (proven invasion of sphincter)
* Diffuse metastatic syndrome (no curative intent, short expected life span)
* preoperative incontinence (non due to the tumor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2001-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Sphincter preservation rate | surgery

SECONDARY OUTCOMES:
Tumor response according to rectal endo-echography | prior to surgery
operative mortality and morbidity | after surgery
anatomopathology margins (lateral and inferior) | after surgery
Functional results (stoma closure, continence, manometry) | 2 years
Local recurrence | 3 years
Disease-free survival | 3 years
Overall Survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rouanet, Pr, Principal Investigator — CRLC Val d'Aurelle
Locations (12):
- France (12):
  - Institut Sainte catherine, Avignon
  - Hopital Saint Andre, Bordeaux
  - Hotel Dieu, Clermont-Ferrand
  - Hopital Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - CAC Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Hopital Saint Eloi, Montpellier
  - Centre Rene Gauducheau, Nantes
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif